CLINICAL TRIAL: NCT02494973
Title: Postoperative Hepatic Arterial Chemotherapy in High-risk Patients as Adjuvant Treatment After Resection of Colorectal Liver Metastases - A Randomized Phase II/III Trial
Brief Title: Postoperative Hepatic Arterial Chemotherapy in High-risk Patients as Adjuvant Treatment After Resection of Colorectal Liver Metastases
Acronym: PACHA-01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-005110-32; 2014/2187 (Other: CSET number)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant systemic chemotherapy with mFOLFOX6 (Active Comparator): started within 8 weeks after surgery for a maximal duration of 6 months and at least 3 months, every 14 days:
  * Oxaliplatin 85 mg/m² in 2 hours IV day (D)1,
  * Acide folinique 400 mg/m² in 2 hours IV (concomitantly to oxaliplatin) D1, followed by 5FU bolus 400 mg/m² in 5-10 minutes IV D1 followed by 5FU 2400 mg/m² IV in 46 hours.
  Interventions: Drug: Oxaliplatin IV; Drug: mFOLFOX6
- Adjuvant HAI oxaliplatin and systemic LV5FU2 (Experimental): started within 8 weeks after surgery for a maximal duration of 6 months and at least 3 months, and performed every 14 days:
  * Oxaliplatin 85 mg/m² in 4-6 hours HAI day (D)1,
  * Acide Folinique 400 mg/m² in 2 hours IV (concomitantly to oxaliplatin) D1, followed by 5FU bolus 400 mg/m² in 5-10 minutes IV D1 followed by 5FU 2400 mg / m² IV in 46 hours. In both arms, continuation of targeted therapy (if any) used in the preoperative treatment is allowed.
  Interventions: Drug: Oxaliplatin HAI; Drug: LV5FU2

INTERVENTIONS:
Drug: Oxaliplatin HAI — Oxaliplatin 85 mg/m² in 2 hours HAI day (D)1,
  Arms: Adjuvant HAI oxaliplatin and systemic LV5FU2
Drug: Oxaliplatin IV — Oxaliplatin 85 mg/m² in 2 hours IV day (D)1,
  Arms: Adjuvant systemic chemotherapy with mFOLFOX6
Drug: mFOLFOX6 — Acide folinique 400 mg/m² in 2 hours IV (concomitantly to oxaliplatin) D1, followed by 5FU bolus 400 mg/m² in 5-10 minutes IV D1 followed by 5FU 2400 mg/m² IV in 46 hours.
  Arms: Adjuvant systemic chemotherapy with mFOLFOX6
Drug: LV5FU2 — Acide Folinique 400 mg/m² in 2 hours IV (concomitantly to oxaliplatin) D1, followed by 5FU bolus 400 mg/m² in 5-10 minutes IV D1 followed by 5FU 2400 mg / m² IV in 46 hours.
  Arms: Adjuvant HAI oxaliplatin and systemic LV5FU2

SUMMARY:
Currently, no adjuvant study with hepatic arterial infusion in the adjuvant setting is opened. Recently, the results of a phase II study (NCT00268463, NSABP-C-09) assessing the potential benefit of systemic oxaliplatin and capecitabine alternating with HAI of FUDR, after resection of CRLM have been reported.

The primary end point was 2-year survival. Fifty-five of 76 eligible patients were able to initiate protocol-directed therapy and completed median of six cycles (range, one to six). Three postoperative or treatment-related deaths were reported. Overall, 88% of evaluable patients were alive at 2 years. With a median followup of 4.8 years, a total of 30 patients have had disease recurrence, 11 involving the liver. Median disease-free survival was 32.7 months. In conclusion alternating HAI of FUDR and systemic capecitabine and oxaliplatin met the prespecified end point of higher than 85% survival at 2 years and were clinically tolerable.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic colorectal adenocarcinoma,
2. Curative-intent resection (or ablation) R0 of at least 4 CRLM,
3. Preoperative oxaliplatin- and/or irinotecan-based chemotherapy (successively or concomitantly) +/- non experimental biological therapy, e.g., anti-EGFR or antiangiogenic antibody,
4. Confirmed radiological tumor control before surgery (i.e., objective response or stable disease according to RECIST1.1 criteria),
5. WHO performance status of 0 or 1,
6. Age ≥ 18 years,
7. Adequate hematological function: absolute neutrophil count (ANC) > 2 x 109/L; platelets > 100 x 10^^9/L, hemoglobin (Hb) > 9 g/dL.
8. Adequate liver function: serum bilirubin </= 1.5 x ULN;
9. Aminotransferases levels </= 2.5 ULN (</= 5 ULN if liver metastases in place), and alkaline phosphatase level ≤ 5 ULN
10. Creatinin clearance ≥ 30 ml/min
11. Informed consent signed by the patient or his/her legal representative.
12. Negative pregnancy test in women of childbearing potential within 14 days prior to treatment initiation (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization). Both men and women (of childbearing potential) who are sexually active must use adequate contraception, during and for at least 6 months post-treatment.

Exclusion Criteria:

1. Extrahepatic metastatic disease (except ≤3 lung nodules (≤10 mm on chest CT scan) deemed amenable to curative-intent resection/ablation),
2. Symptomatic primary tumor requiring urgent surgery, asymptomatic primary colorectal tumor is not a non-inclusion criteria if its
3. Contraindication to fluoropyrimidines or oxaliplatin, as mentioned in the SMPC of investigational medicinal products
4. Known dihydropyrimidine dehydrogenase (DPD) deficiency
5. Disease progression during, or early hepatic relapse (< 6 months) after the end of, oxaliplatin-based adjuvant chemotherapy following primary tumor resection
6. History of hepatic arterial infusion with any treatment (chemotherapy, radioembolisation),
7. Peripheral neuropathy> grade 1,
8. History of cancer within 5 years prior to entry into the trial other than adequately treated basal-cell skin cancer or in situ carcinoma of the cervix
9. Concomitant administration of cimetidine
10. Concomitant medications/comorbidities that may prevent the patient from receiving study treatments,
11. Patient already included in another clinical trial with an experimental molecule,
12. Pregnancy or lactation,
13. Patients deprived of liberty or under guardianship,
14. Patients unable to undergo medical monitoring test for geographical, social or psychological reasons.
15. Patients must not have any uncontrolled concurrent illness including, but not limited to, severe active or uncontrolled infection, symptomatic congestive heart failure, unstable, angina pectoris, cardiac arrhythmia, uncontrolled diabetes mellitus or psychiatric illness/social situations that would limit compliance with study requirements resection is planned (REVERSE strategy authorized)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
18-month hepatic RFS rate | Assessed 18 months after inclusion
3-year RFS rate | Assessed 3 years after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Goere D, Pignon JP, Gelli M, Elias D, Benhaim L, Deschamps F, Caramella C, Boige V, Ducreux M, de Baere T, Malka D. Postoperative hepatic arterial chemotherapy in high-risk patients as adjuvant treatment after resection of colorectal liver metastases - a randomized phase II/III trial - PACHA-01 (NCT02494973). BMC Cancer. 2018 Aug 6;18(1):787. doi: 10.1186/s12885-018-4697-7. PMID 30081865